CLINICAL TRIAL: NCT04083690
Title: Multi-lead ECG to Effectively Optimize Resynchronization Devices: New CRT Recipients
Acronym: METEOR-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Alan J. Bank, MD, Medical Director of Research - United Heart & Vascular Clinic, Allina Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRBnet#: 1455594
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Systolic
Keywords: Cardiac Resynchronization Therapy; Pacing; Echocardiography; Electrocardiography; Optimization; Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: 1:1 randomization - active comparator and experimental arm (note: at 6 months the control arm will crossover)
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients blinded to which study group they randomized and how their CRT device is programmed. Individuals (readers) who perform echocardiographic measurements blinded to patient randomization and CRT settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard CRT Programming, then ECG CRT Optimization (Active Comparator): The control arm patients will have standard CRT programming for the first 6 months, and then will be reprogrammed based on the ECG CRT optimization information for the following 6 months
  Interventions: Device: Reprogramming of CRT Device Settings to Optimal Electrical Synchrony
- ECG CRT Optimization (Experimental): The experimental arm patients will have CRT device reprogrammed based on the ECG CRT optimization information for 12 months.
  Interventions: Device: Reprogramming of CRT Device Settings to Optimal Electrical Synchrony

INTERVENTIONS:
Device: Reprogramming of CRT Device Settings to Optimal Electrical Synchrony — Reprogramming of CRT device to maximize the benefit based on the ECG CRT optimization information.

SUMMARY:
Cardiac resynchronization therapy (CRT), or atrial-synchronized biventricular (BiV) pacing, is an FDA-approved device therapy option for heart failure (HF) patients with reduced left ventricular ejection fraction and electrical dyssynchrony. A traditional CRT device has pacing leads implanted within the right atrium (RA), the right ventricle (RV), and within a coronary vein overlying the lateral or posterior left ventricle (LV). Within the past decade, various multi-center randomized controlled trials have reported improved quality of life, aerobic exercise capacity, LV systolic function and structure, as well as decreased hospitalization rates and mortality among patients with HF. Despite improvements in CRT technology with multipoint pacing, quadripolar leads, and adaptive pacing algorithms, approximately 30% of patients do not clinically benefit and are considered non-responders. This study looks to optimize new CRT device recipients using information obtained from standard ECG machines.

DETAILED DESCRIPTION:
This is a prospective, randomized study designed to evaluate if CRT device optimization, guided by electrocardiography, improves echocardiographic and clinical outcomes among HF patients with a CRT device implanted for standard indications. All patients will have measurement of electrocardiograms at a range of device settings. Patients will be randomized in a 1:1 ratio to either the active comparator arm (standard CRT programming), or the experimental arm (CRT device programmed by the information obtained by ECGs). Standard CRT programming used in this study is simultaneous biventricular (BiV) pacing with a fixed atrioventricular delay. At 6 months, control patients who were initially randomized to standard programming will have programming changed based on the ECG optimization information. Patients will be blinded to randomization. Change of LV size and function will be performed prior to randomization, and again ~6 and ~12 months following CRT implant in both subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (or their legal guardian) must be willing to provide informed consent and sign a data privacy authorization (HIPAA) form
2. Age greater than or equal 18 years
3. Pre-CRT EF less than or equal 40%
4. Patients will be receiving or have received a first-time CRT device for standard clinical indications within ~2 months of study enrollment
5. Adequate echocardiographic images for LV EF and LV ESV determination
6. On optimal medical therapy

Exclusion Criteria:

1. Patients who are pregnant or may become pregnant
2. Patient has a history of severe allergic reactions from ECG gel/ electrode adhesives
3. Patient has a His Bundle pacing lead
4. Patient has right bundle branch block (RBBB)
5. Patient is enrolled in concurrent research study that would potentially confound the results of this study
6. Premature ventricular contraction (PVC) burden greater than or equal to 10%

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular size | 6 months
  Change in left ventricular end-systolic volume (LVESV), measured by echocardiogram, in patients in the experimental arm vs active comparator arm

SECONDARY OUTCOMES:
Change in left ventricular function | 6 months
  Change left ventricular ejection fraction (EF), measured by echocardiogram, in patients in the experimental arm vs active comparator arm
Change in left ventricular size | 6 months
  Change in LVESV, measured by echocardiogram, in the subset of patients with left bundle branch block (LBBB) or intraventricular conduction delay (IVCD) in the experimental arm vs the active comparator arm
Change in left ventricular size | 6 months
  Change in LVESV, measured by echocardiogram, in the subset of patients with complete heart block (CHB) or persistent atrial fibrillation (AF) in the experimental arm vs the active comparator arm
Change in left ventricular size | 6 months
  Change in LVESV, measured by echocardiogram, in patients in the active comparator arm (crossed-over to optimization device settings at 6 months) at 12 months vs 6 months

OTHER OUTCOMES:
Correlation of change in electrical dyssynchrony and LVESV | 12 months
  Changes in electrical dyssynchrony, as measured by electrocardiography (ECG) and correlation to change LVESV, measured by echocardiogram, in the entire patient cohort

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, MD, Principal Investigator — United Heart & Vascular - Allina Health System
Locations (2):
- United States (2):
  - Minneapolis Heart Institute (Abbott Northwestern Hospital), Minneapolis, Minnesota
  - United Heart & Vascular Clinic, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers